

| Participant Study ID: |
|-----------------------|
| antioipaint otalaj ib |

## **CONSENT FORM**

Study title: The Role Of Virtual Dietetic Interventions In Patients With Coeliac Disease

Name of Researcher: [insert CI name]

Please initial box

| 1 | I confirm that I have read the<br>the above study. I have had t<br>questions and have had these | the opportunity to con | sider the information, ask |
|---|---|---|---|
| 2 | I understand that my participa<br>at any time without giving any<br>being affected. | • | |
| 3 | I understand that participation involves receiving pre-recorded educational advice in relation to the gluten-free diet for coeliac disease from a gastroenterology dietitian. If I am allocated to this group of participants; I understand that I will not receive the normal initial consultation with the dietician – just the follow up session. | | |
| 4 | I understand that researchers from my direct care team may also use de-<br>identified clinical data from my medical records to during this research. | | |
| 5 | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records to make sure the research has been managed correctly. | | |
| 6 | I agree to take part in the above study | | |
| 7 | OPTIONAL: I agree that data collected for this study can be used for future research and may be shared anonymously with external researchers based worldwide, as detailed in the information sheet. | | |
| Na | ime of Participant | Date | Signature |
| Na | me of Person taking consent | Date | Signature |

When completed: 1 for participant; 1 for researcher site file; 1 (original) to be kept in medical notes.